CLINICAL TRIAL: NCT03354299
Title: Beneficial Effects of Coconut Milk Supplementation to Improve Nutritional Status in Patients With Liver Cirrhosis
Brief Title: Effect of Coconut Milk Supplementation to Improve Nutritional Status in Cirrhosis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Rino Alvani Gani, Head of Hepatobiliary, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 75/UN2.F1/ETIK/2015
Record Dates: First submitted 2017-11-13; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Malnutrition; Cirrhosis, Liver
Keywords: malnutrition; liver cirrhosis; coconut milk
MeSH Terms: conditions — Malnutrition; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: The patients were divided into 2 groups, groups I received 25 g of sugar plus 50 cc of coconut milk (200 kkal) as late night snacks (LNS); and group II received 50 g of sugar alone (200 kkal) as LNS

ARMS (2):
- Group I (Experimental): Group I patients received 25 gram of sugar (pudding) and 50 cc of coconut milk as late night snack for a month
  Interventions: Dietary Supplement: coconut milk
- Group II (Active Comparator): Group II patients received 50 gram of sugar (25 gram pudding and 25 gram syrup) as late night snack for a month
  Interventions: Dietary Supplement: coconut milk

INTERVENTIONS:
Dietary Supplement: coconut milk — 50 cc of coconut milk supplementation plus 25 gram sugar (pudding) was given to cirrhosis patients as late night snack

SUMMARY:
Liver cirrhosis still becomes a major issue in Indonesia. Malnutrition has been observed in liver cirrhosis patients as it deteriorates liver function and cirrhosis itself. Malnutrition in liver cirrhosis can increase morbidity and mortality rates.

Patients with liver cirrhosis have increased energy expenditure and endogenous fat oxidation reaction which is used as the basic energy sources. Energy obtained from fat was accounted for 86% of the total energy sources in this population. Fatty acid is also known to be an efficient energy backup for hepatocytes and other cells because it generates higher adenosine triphosphate (ATP) than other sources.

Supplementary diet for patients with liver cirrhosis is considered beneficial for preventing hypercatabolism. To fulfill their nutritional needs, patients with liver cirrhosis is advised to take an extra food, such as a late night snack (LNS) with a total carbohydrate of around 50 g (equivalent to 200 kkal). Considering that most of the energy source in patients with liver cirrhosis came from fat, so the additional sources of energy having a high fat content were considered to be potentially highly beneficial to address the patients' nutritional status, as well as to reduce the risk of hyperglycemia after a meal and hypoglycemia after a long night fasting period time.

Coconut milk contains many saturated fatty acids belonging to the medium chain triacylglycerol (MCT) group. The characteristics of MCT are quite different from long chain triacylglycerol (LCT). MCTs are more easily absorbed than LCTs, and are mostly absorbed in the form of free fatty acids, in both healthy and liver cirrhosis populations.

This study wants to investigate the effects of coconut milk supplementation on improving the nutritional status of patients with liver cirrhosis. The patients were divided into 2 groups, groups I received 25 g of sugar plus 50 cc of coconut milk (200 kkal) as late night snacks (LNS); and group II received 50 g of sugar alone (200 kkal) as LNS. Investigators think that the group who received coconut milk supplementation has better nutritional status than the other group.

DETAILED DESCRIPTION:
This study investigated the effects of coconut milk supplementation on improving the nutritional status of patients with liver cirrhosis. Design was randomized controlled trial. Investigators randomized the patients into 2 groups. Group I received 25 gram of sugar + 50 cc coconut milk and group II received 50 gram of sugar alone. Both of groups received 200 kkal as late night snack. Subjects were cirrhosis patients with Child Pugh A and B, who develop malnutrition using BMI criteria or experience unintentional weight loss. The outcome was nutritional parameters after 1 month supplementation.

Estimated sample was 60 patients with 30 subjects in group I and 30 subjects in group II.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis patients, Child Pugh A and B who are not critically ill, and develop one of following condition :

  1. Malnutrition with modified BMI criteria such as BMI < 22 kg/m2 for non ascites, BMI < 23 for mild ascites, and BMI < 25 for severe ascites
  2. Unintentional weight loss, defined as decline 5% weight loss for period 6-12 month or less

Exclusion Criteria:

* Using pace maker
* Diabetes mellitus patients
* End-stage renal disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Change of BMI at 1 month after supplementation
  Body mass index is calculated by divided weight (in kg) with square of height (in meter). Unit of measure: kg/m2
Triceps Skinfold Thickness (TSF) | Change of TSF at 1 month after supplementation
  Triceps skinfold thickness is calculated by skinfold calliper. Unit of measure: millimeter (mm)
MAMC (Mid arm muscle circumference) | Change of MAMC at 1 month after supplementation
  Mid arm muscle circumference is calculate by formula as follow:
  MAMC = MUAC - (TSF x 3.14). MUAC (mid upper arm circumference). Unit of measure: milimeter (mm)
Body Fat Mass (BFM) | Change of BFM at 1 month after supplementation
  Body fat mass is calculated by calliper by pulling the fat away from the muscles, pinch them with the caliper, take the measurements, and look at a chart to figure out. Unit of measure : kg
Prealbumin and albumin serum | Change of prealbumin and albumin serum at 1 month after supplementation
  Prealbumin serum is checked by nephelometry technique with nephelometer laser, albumin serum is checked by bromcresol green method, using ABX cobas. Both of that in milligram per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Rino A Gani, PhD, Principal Investigator — Dr
Locations (1):
- Hepatobiliary Division, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided